CLINICAL TRIAL: NCT06040996
Title: A Randomized Controlled Trial of Improving Parenting Skills Adult ADHD (IPSA): A New Parent Training Program for Parents Who Themselves Have ADHD
Brief Title: Evaluation of Improving Parenting Skills Adult ADHD (IPSA): A New Parent Training Program for Parents With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPSA RCT
Record Dates: First submitted 2023-08-28; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Parenting; Adult ADHD; Parent-Child Relations; Child Behavior Problem
Keywords: Parenting; Parent training; Parental ADHD; Parenting skills; Parental Self-Efficacy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPSA (Experimental): A new parent training program for parents with ADHD
  Interventions: Behavioral: Improving Parenting Skills adult ADHD (IPSA)
- Continued Routine Services (Other): Continued Routine Services
  Interventions: Other: Continued Routine Services

INTERVENTIONS:
Behavioral: Improving Parenting Skills adult ADHD (IPSA) — Parent training program for parents with ADHD. The program combines structured group-based skills training with individualized support, including occupational therapist support to help parents improve their own prerequisites for bringing about change and facilitate use of the introduced parenting skills.
  Arms: IPSA
Other: Continued Routine Services — Continued Routine Services while waiting for IPSA (offered approximately 6 months later)
  Arms: Continued Routine Services

SUMMARY:
IPSA (Improving Parenting Skills adult ADHD) is a new parent training (PT) program developed and adapted for parents who themselves have Attention-Deficit/Hyperactivity Disorder (ADHD).

This study evaluates the efficacy of the IPSA program, that is, whether participation in IPSA is associated with desired treatment outcomes (e.g., improved parental self-efficacy). In addition, it examines the program's feasibility (e.g., what parents think about the program, the extent to which parents complete the program, and program safety).

The study is a so called randomized controlled trial (RCT), where participants are randomly assigned to one of two groups: Treatment (IPSA) or Control (continued routine services; offered IPSA approximately six months later).

Participants are adults with ADHD (any form) that have at least one child in the ages between 3 and 11 years. Data are primarily collected using questionnaires, completed by parents before and after IPSA, as well as in connection with an IPSA booster session (follow-up).

DETAILED DESCRIPTION:
DESIGN: An RCT with parallel groups, where eligible individuals are block randomized on each clinical site to one of two groups (ratio 1:1): Treatment (IPSA directly) or Control (continued routine services; offered IPSA approximately six months later). Each block includes 18 participants. Randomization is done using a digital randomization tool. Allocation (treatment or control) is masked to participants and study staff administering the screening/inclusion/assessment procedures until after the baseline assessment (including pre-intervention questionnaires) has been completed.

SETTING: The study is carried out by the Center of Neurodevelopmental Disorders at Karolinska Institutet (KIND), Karolinska Institutet, Sweden, in collaboration with an ADHD Center run by the publicly-funded Habilitation & Health, Stockholm Health Care Services, Region Stockholm, Sweden. Originally, the plan was to gradually involve external clinical sites (e.g., regular outpatient psychiatric clinics) in the data collection. However, this plan was first postponed and later cancelled due to the Covid-19 pandemic.

ETHICS: The study has been approved by the Regional Ethics Committee of Stockholm, Sweden (dnr. 2017/2435-31/5, 2019-06362, and 2023-03871-02).

PARTICIPANTS: Parents (≥ 18 years of age) with a formal ADHD diagnosis (any form) having at least one child aged 3 to 11 years, recruited via the project web site as well as among families enrolled at the involved clinical site.

SAMPLE SIZE: Power calculations (with 1 - β = .80, α = .05, medium to large effect sizes) has resulted in an estimated sample size of n ≥ 100.

RESEARCH QUESTIONS: The research questions are primarily concerned with the efficacy of IPSA, secondarily with the feasibility of the program. In addition, the investigators will explore the potentially moderating or mediating effects of baseline variables and levels of active participation on efficacy outcomes.

EFFICACY: The effect of IPSA is examined using self- and parental report scales administered before (pre; T1) and immediately after (post; T2) IPSA, as well as approximately 1.5-3 months after program completion, in connection with an IPSA booster session (follow-up; T3). Specifically, the investigators examine whether participation in IPSA is associated with positive treatment outcomes with respect to the study's primary outcome (parental self-efficacy) and secondary outcomes (parental stress, levels of household disorganization or frequency and perception of disruptive behavior problems in the participant's target child). In addition, parents' time management and organizational skills are followed from pre to post IPSA.

FEASIBILITY: The feasibility of IPSA is evaluated based attendance records and parental reports. The investigators assess whether IPSA is an acceptable intervention (i.e., treatment satisfaction, treatment credibility), examine levels of active participation (i.e., program completion rates, levels of homework completion, use of introduced parenting skills, and management of a targeted parent-child interaction situation), and monitor potential harms (including parental reports of general perceived stress, symptoms of anxiety/depression and adverse events).

TREATMENT INTEGRITY: Intervention sessions are recorded (audio only). Treatment integrity (assessed in terms of facilitator adherence/fidelity) is examined in 20% of group sessions (randomly selected), using checklists covering program elements and content.

ELIGIBILITY:
Inclusion Criteria: Adults (≥ 18 years) with a formal ADHD diagnosis (any form), having:

* at least one child in the ages between 3 and 11 years
* sufficient knowledge of Swedish to participate actively in the intervention without an interpreter
* possibility to participate in the intervention during the intended period (regardless of allocation)

Exclusion Criteria:

* other neurodevelopmental disabilities, that is autism or intellectual disability
* ongoing serious psychiatric condition (e.g., major depression, suicidality, psychosis, substance use disorder) for which treatment needs to be prioritized
* ongoing family crisis or equivalent that needs to be prioritized with other types of interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Parental Self-Efficacy | Administered at baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the Parental Self-Efficacy scale (PSE; Ulfsdotter, Enebrink, & Lindberg, 2014). Expected to change from pre to post IPSA. Higher scores mean better outcome.

SECONDARY OUTCOMES:
Parental Stress | Administered at baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the Parental Stress Scale (PSS; Berry & Jones, 1995). Assessed for change from pre to post IPSA. Lower scores mean better outcome.
Household Disorganization/Home Chaos | Administered at baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the Confusion, Hubbub, and Order Scale (CHAOS; Matheny, Wachs, Ludwig, & Phillips, 1995). Assessed for change from pre to post IPSA. Lower scores mean better outcome.
Child behavior problems | Administered at baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the Eyberg Child Behavior Inventory (ECBI; Axberg, Johansson Hanse, & Broberg, 2008; Eyberg & Ross, 1978). Assessed for change from pre to post IPSA. Lower scores mean better outcome.

OTHER OUTCOMES:
Time management and organizational skills | Administered at baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2).
  Measured with the Swedish Assessment of Time Management Skills (ATMS-S; Roshanay, Janeslätt, Lidström-Holmqvist, White, & Holmefur, 2022). Assessed for change from pre to post IPSA. Higher scores mean better outcome.
Feasibility (acceptability): Program acceptability | Immediately after program completion (up to six months after baseline).
  Overall treatment satisfaction (i.e., satisfaction with the IPSA program as a whole) is assessed with a treatment evaluation questionnaire (Bramham et al., 2009) modified to fit the PT context. A summary mean score of ≥ 3 (out of 4) is interpreted as a positive evaluation, indicating satisfactory acceptability. In addition, the scale has been supplemented with a summative grade for the program (mimicking school grades fail, pass, pass with distinction, and pass with special distinction), a question about the likelihood of the parent recommending IPSA to others, and two open-ended questions about how IPSA has been good/helpful or could be made better/more helpful.
Feasibility (acceptability): Session acceptability | At the end of each IPSA session, up to the booster session (up to three months after program completion).
  Treatment satisfaction with separate IPSA sessions is measured using a subset of questions from a treatment evaluation questionnaire (Bramham et al., 2009), modified to fit the PT context. A summary mean score of ≥ 3 (out of 4) is interpreted as satisfactory positive.
Feasibility (acceptability): Intervention Credibility | Up to six weeks after baseline.
  Assessed using the Credibility/Expectancy Questionnaire (C/EQ; Devilly & Borkovec, 2000), modified to fit the PT context. Higher ratings indicate more/higher credibility.
Feasibility (active participation): Program completion | Attendance is registered for every IPSA session, up to the booster session (up to three months after program completion).
  Program completion rates are assessed based on the percentage of program starters who attend at least nine of the 14 regular IPSA sessions. For us to say that treatment completion is good, we want at least 75 % of participants to have completed the program.
Feasibility (active participation): Homework completion | At the beginning of IPSA sessions 6 through 14 (up to six months after baseline).
  Assessed using the first two items of the Homework Rating Scale (Kazantzis, Deane, & Ronan, 2004), adapted to the PT context. Higher ratings indicate greater homework completion quantity or quality, respectively.
Feasibility (active participation): Use of introduced parenting skills | At baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Participants' use of parenting skills addressed during IPSA is measured with 11 questions about the frequency of targeted parental behaviors and activities. Higher scores mean better outcome.
Feasibility (active participation): Management of a targeted parent-child interaction situation | During the first and the last regular IPSA sessions (up to six months after baseline).
  As part of the IPSA program's follow-up procedures, participants rate their performance in managing an individually defined "IPSA situation" (on a scale from 0 = not at all good - 10 = very good) as well as their satisfaction with their way of managing their "IPSA situation" (on a scale from 0 = not at all satisfied to 10 = very satisfied). Higher scores mean better outcome.
Feasibility (potential harms): General perceived stress | At baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the 10-item version of the Perceived Stress Scale (PSS-10; Cohen, Kamarck, & Mermelstein, 1983; Nordin & Nordin, 2013). Lower scores mean better outcome.
Feasibility (potential harms): Anxiety/Depression | At baseline (pre IPSA; T1) and immediately after the intervention (post IPSA; T2), as well as at follow-up (up to three months after program completion; T3).
  Measured with the Hospital Anxiety and Depression Scale (HADS; Lisspers, Nygren, & Söderman, 1997; Zigmond & Snaith, 1983). Lower scores mean better outcome.
Feasibility (potential harms): Adverse Events and Serious Adverse Events | Up to the follow-up (up to three months after program completion).
  Monitored by documenting spontaneously reported adverse events (e.g., any unfavorable, potentially negative, event that occur during the study period) and serious adverse events (e.g., threatening life or function; requiring hospitalization).

CONTACTS AND LOCATIONS:
Overall Officials: Tatja Hirvikoski, Ass. Prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Lindstrom T, Buddgard S, Westholm L, Forster M, Bolte S, Hirvikoski T. Parent training tailored for parents with ADHD: a randomized controlled trial. BMC Psychiatry. 2025 Aug 26;25(1):818. doi: 10.1186/s12888-025-07166-8. PMID 40859158